CLINICAL TRIAL: NCT02189122
Title: Comparative Effects of Rapid-Release Aspirin and NHP-544C on Basal and Bradykinin Stimulated Prostacyclin Production
Brief Title: Comparative Effects of Aspirin and NHP-544C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Nancy J. Brown, M.D.; Professor of Medicine and Pharmacology, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 140707
Record Dates: First submitted 2014-07-10; First posted 2014-07-14 (Estimated); Results first posted 2016-06-03 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
MeSH Terms: interventions — Bradykinin; Aspirin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1:Aspirin/placebo (Active Comparator): Group 1 will be randomized to the order in which they receive rapid-release aspirin (ASA), 81 mg), ASA 162.5 mg, and identical-appearing placebo for 5 days. Bradykinin will be given intravenously in graded doses on the fifth day of each treatment period.
  Interventions: Drug: Bradykinin; Drug: Aspirin 81 mg; Drug: Aspirin 162 mg; Drug: Placebo
- Group 2:NHP-544C/placebo (Active Comparator): Group 2 will be randomized to the order in which they receive NHP-544C 81 mg, NPH-544C 162.5 mg and identical-appearing placebo for five days. Bradykinin will be given intravenously in graded doses on the fifth day of each treatment period.
  Interventions: Drug: Bradykinin; Drug: NHP544-C 81 mg; Drug: NHP544C 162 mg; Drug: Placebo

INTERVENTIONS:
Drug: Bradykinin — Bradykinin will be given intravenously in graded doses. Each dose will be given for 15 minutes.
  Other Names: BK
Drug: Aspirin 81 mg — Subjects will take Aspirin 81 mg per day for five days.
  Other Names: ASA 81 mg
  Arms: Group 1:Aspirin/placebo
Drug: Aspirin 162 mg — Subjects will take aspirin 162 mg per day for 5 days.
  Other Names: ASA 162 mg
  Arms: Group 1:Aspirin/placebo
Drug: NHP544-C 81 mg — Subjects will take NHP544C 81 mg per day for five days.
  Arms: Group 2:NHP-544C/placebo
Drug: NHP544C 162 mg — Subjects will take NHP544C 162 mg once a day for five days.
  Arms: Group 2:NHP-544C/placebo
Drug: Placebo — Subjects will take matching placebo for five days.

SUMMARY:
The investigators will compare the effects of rapid release aspirin and NHP-544C on the prostacyclin response to intravenous bradykinin.

ELIGIBILITY:
Inclusion Criteria:

1. Ages of 18 and 55 years, inclusive
2. No significant medical issues without significant abnormal findings at the baseline physical examination
3. Body mass index (BMI) between 18.0 and 30.0kg/m2 (weight (kg)/[height(m)]2)
4. For women - negative pregnancy test on Period 1, Day -1, or surgically sterilized, or is at least two years post-menopausal prior to randomization. Females of childbearing potential must be practicing an acceptable method of birth control to be eligible. Acceptable forms of birth control include: condom plus spermicide or condom plus other form of birth control including hormonal method (IUD, patch, ring, implant, or injectable), sterilization of partner, or non-hormonal IUD. The use of oral contraceptives is allowed during the study, but the subject must be on a stable dose for 30 days prior to the trial and throughout all four dosing periods
5. Ability to understand the requirements of the study and a willingness to comply with all study procedures

Exclusion Criteria:

1. Clinically significant and relevant medical history (including failure of a major organ system) or current medical illness, and is deemed by the Principal Investigator to be unsuitable to participate in the study
2. Participation in an investigational drug study within the 30 days prior to CRC admission
3. Use of aspirin or other NSAID within 14 days of Day 1 of the study. All other medications, prescription (with the exception of contraceptives), over-the-counter (OTC), herbal, and vitamin supplements must be discontinued 7 days prior to Day 1. If subjects are taking prescription medication, or OTC medication at the direction of a health care provider, that provider must confirm that it is acceptable for them to stop dosing for the duration of the study
4. History of metabolic, renal, hepatic, hemorrhagic stroke, gastrointestinal bleed, cardiovascular disease, central nervous system disorder, or peptic ulcer disease or other chronic bleeding disorder
5. History of gastrointestinal disorder that could result in incomplete absorption of the study drug
6. Malignancy, or neurologic or psychiatric disorder
7. Abnormal laboratory value(s) determined to be clinically significant (in the opinion of the Investigator)
8. History of illicit drug abuse in the past year or current evidence of such abuse in the opinion of the investigator
9. Pregnancy or lactation
10. Acute illness within 1 week of CRC admission
11. Significant loss of blood or blood or plasma donation within 30 days of drug administration
12. Hypersensitivity or allergy to NSAIDs, aspirin, ethylcellulose, polyvidone, castor oil, magnesium stearate, tartaric acid, colloidal anhydrous silica, talc, gelatin, titanium dioxide, erythrosine, or indigotin
13. History of aspirin resistance
14. History of alcohol abuse within past year. Current alcohol use should not exceed 14 standard alcoholic drinks per week. A drink is defined as 1.5 ounces (oz.) liquor, 12 oz. beer, or 6 oz. wine
15. Alcohol consumption within 3 days of Day 1
16. Difficulty swallowing oral medications
17. Consumption of coffee or caffeine-containing beverages exceeding the equivalent of five 8-oz cups of coffee per day on average

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy J Brown, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Gamboa JL, Devin JK, Ramirez CE, Yu C, Nian H, Lee RH, Brown NJ. Comparative effects of immediate-release and extended-release aspirin on basal and bradykinin-stimulated excretion of thromboxane and prostacyclin metabolites. Pharmacol Res Perspect. 2016 Feb 23;4(2):e00221. doi: 10.1002/prp2.221. eCollection 2016 Apr. PMID 27069632

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-five enrolled participants were excluded prior to randomization to study group because they did not meet inclusion or exclusion criteria.
Groups:
- Group 1:Aspirin/Placebo: Group 1 will be randomized to receive rapid release aspirin (ASA, 81 mg), ASA 162.5 mg, or identical-appearing placebo for 5 days. Bradykinin will be given intravenously in graded doses on the fifth day of study.
  Bradykinin: Bradykinin will be given intravenously in graded doses. Each dose will be given for 15 minutes.
  Aspirin 81 mg: Subjects will take Aspirin 81 mg per day for five days.
  Aspirin 162 mg: Subjects will take aspirin 162 mg per day for 5 days.
  Placebo: Subjects will take matching placebo for five days.
  Three subjects participated in each possible sequence with the following exceptions: Four subjects participated in the sequence Aspirin 81 mg, Aspirin 162.5 mg, placebo; two subjects participated in the sequence placebo, Aspirin 162.5 mg, Aspirin 81 mg.
- Group 2:NHP-544C/Placebo: Group 2 will be randomized to receive NHP-544C 81 mg, NPH-544C 162.5 mg or placebo. Bradykinin will be given intravenously in graded doses on the fifth day of study drug.
  Bradykinin: Bradykinin will be given intravenously in graded doses. Each dose will be given for 15 minutes.
  NHP544-C 81 mg: Subjects will take NHP544C 81 mg per day for five days.
  NHP544C 162 mg: Subjects will take NHP544C 162 mg once a day for five days.
  Placebo: Subjects will take matching placebo for five days.
  Three subjects participated in each possible sequence with the following exceptions: Four subjects participated in the sequence NHP544C 81 mg, NHP544C 162 mg, placebo; two subjects participated in the sequence NHP544C 162 mg, placebo, NHP544C 81 mg.
Period: Overall Study
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1:Aspirin/Placebo: Group 1 will be randomized to receive rapid release aspirin (ASA, 81 mg), ASA 162.5 mg, or identical-appearing placebo for 5 days. Bradykinin will be given intravenously in graded doses on the fifth day of study.
  Bradykinin: Bradykinin will be given intravenously in graded doses. Each dose will be given for 15 minutes.
  Aspirin 81 mg: Subjects will take Aspirin 81 mg per day for five days.
  Aspirin 162 mg: Subjects will take aspirin 162 mg per day for 5 days.
  Placebo: Subjects will take matching placebo for five days.
- Group 2:NHP-544C/Placebo: Group 2 will be randomized to receive NHP-544C 81 mg, NPH-544C 162.5 mg or placebo. Bradykinin will be given intravenously in graded doses on the fifth day of study drug.
  Bradykinin: Bradykinin will be given intravenously in graded doses. Each dose will be given for 15 minutes.
  NHP544-C 81 mg: Subjects will take NHP544C 81 mg per day for five days.
  NHP544C 162 mg: Subjects will take NHP544C 162 mg once a day for five days.
  Placebo: Subjects will take matching placebo for five days.
- Total: Total of all reporting groups
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Continuous [Mean (Inter-Quartile Range); unit: years] | 27.4 [24.2 to 33.6] | 26.5 [24.1 to 28.4] | 27.1 [24.1 to 33.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 13 | 21
  Male | 10 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 15 | 17 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 18 | 14 | 32
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
11-dehydrothromboxane B2 [Median (Inter-Quartile Range); unit: ng/mg creatinine] | 0.180 [0.158 to .240] | .214 [.191 to .296] | .206 [.172 to .272]
2,3-dinor-6-keto-PGF1alpha [Median (Inter-Quartile Range); unit: ng/mg creatinine] | .1 [.089 to .139] | .139 [.117 to .252] | .121 [.095 to .158]

OUTCOME MEASURES:

1. Primary Outcome: Urine Thromboxane Concentrations at Placebo ASA or Placebo NHP-544C Dose
Time Frame: 24 hour collection
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Number analyzed (Participants) | 18 | 18
ng/mg creatinine | 0.181 [0.143 to 0.216] | 0.255 [0.219 to 0.322]

2. Primary Outcome: Urine Thromboxane Concentrations at 81mg ASA or NHP-544C Dose
Time Frame: 24 hour collection
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Number analyzed (Participants) | 18 | 18
ng/mg creatinine | 0.0685 [0.0585 to 0.0717] | 0.115 [0.095 to 0.155]

3. Primary Outcome: Urine Thromboxane Concentrations at 162.5 mg ASA or NHP-544C Dose
Time Frame: 24 hour collection
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Number analyzed (Participants) | 18 | 18
ng/mg creatinine | 0.054 [0.043 to 0.077] | 0.071 [0.056 to 0.115]

4. Primary Outcome: Urine Prostacyclin Concentrations at Placebo ASA or Placebo NHP-544C Dose
Time Frame: 24 hour collection
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Number analyzed (Participants) | 18 | 18
ng/mg creatinine | 0.102 [0.083 to 0.116] | 0.144 [0.128 to 0.194]

5. Primary Outcome: Urine Prostacyclin Concentrations at 81 mg ASA or NHP-544C Dose
Time Frame: 24 hour collection
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Number analyzed (Participants) | 18 | 18
ng/mg creatinine | 0.069 [0.049 to 0.116] | 0.128 [0.105 to 0.161]

6. Primary Outcome: Urine Prostacyclin Concentrations at 162.5 mg ASA or NHP-544C Dose
Time Frame: 24 hour collection
Population: Data are given for 162.5 mg study day
Measure: Median (Inter-Quartile Range); unit: ng/mg creatinine
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Number analyzed (Participants) | 18 | 18
ng/mg creatinine | 0.067 [0.045 to 0.104] | 0.108 [0.084 to 0.160]

ADVERSE EVENTS:
Arm/Group | Group 1:Aspirin/Placebo | Group 2:NHP-544C/Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 7/18 | 6/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1:Aspirin/Placebo (N=18) | Group 2:NHP-544C/Placebo (N=18)
ST T wave changes following bradykinin infusion (Cardiac disorders) | 2 (2) | 3 (3)
Sinus or nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
low albumin (Hepatobiliary disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes